CLINICAL TRIAL: NCT05960903
Title: Patient Satisfaction After Primary Total Hip Arthroplasty In Assiut University Hospitals
Brief Title: Patient Satisfaction After Primary THA In Assiut University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hamza Sayed Mohamed, Doctor, Assiut University
Other Study IDs: Satisfaction in (THA)
Record Dates: First submitted 2023-06-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
measure the level of patient satisfaction after THA at the arthroplasty unit of Assiut University Hospital.

DETAILED DESCRIPTION:
A dedicated sheet will be used to record patients' data including all demographic data, detailed analysis of time of injury, time and details of surgery . Investigators conduct retrospective study and review the case detalis for 50 eligible patients who underwent total hip arthroplasty between December 2021 and December 2022 in our Assiut University Orthopaedics and Trauma surgery Department All patients followed and evaluated in our outpatient clinic at 3 month post-operatively. In addition to clinical, neurological, and radiological examination, a dedicated and validated questionnaire will be used for measuring the clinical and functional outcome at each visit.

The questionnaire includes three majors parts (1) general satisfaction level after total hip arthroplasty .(2) satisfaction level for 16 subordinate items : pain relief, walking on a flat surface , ascending stairs , getting in/out of cars, squatting, rising after squatting, putting on and tying shoes, walking fast or jogging, limp length discrepancy , hip squeaking( cases of ceramic and non ceramic implant) , hip stiffness, abnormal feeling in the hip, muscle weakness when walking, hip numbness and discomfort in cold weather(3) Ranking the top 5 important functions or issues among the 16 items , with "important" being defined as what patients are currently most concerned with.Objective The Harris Hip Scale (HHS) was developed for the assessment of the results of hip surgery such as total hip arthroplasty , and we intended to use it in evaluation of patient satisfaction level There are ten items covering four domains. The domains are pain, function, absence of deformity, and range of motion The pain domain measures pain severity and its effect on activities and need for pain medication. The function domain is divided into daily activities and gait. The deformity domains observes hip flexion, adduction, internal rotation, and extremity length discrepancy while the range of motion domain asses hip (ROM) .The Harris Hip Score (HHS) is divided into three sections. The first section are questions about pain and its impact which are answered by the patient or client. The second and third sections require the clinician The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible is 100. Results can be interpreted with the following <70 = very dissatisfied result; 70-80 = somewhat dissatisfied , 80-90 = somewhat satisfied , and 90-100 = very satisfied .then a two category satisfaction outcome was determined for each question by combining patients who answered very dissatisfied , dissatisfied into " Dissatisfied group " and combining those who answered satisfied or very satisfied into " Satisfied group " . These two categories were used for all statical analysis

The Oxford Hip Score (OHS) is a joint-specific, patient-reported outcome measure designed to assess disability in patients undergoing total hip arthroplasty Its' primary goal during development was to assess pain and function in patients undergoing joint replacement surgery.

The OHS is a short 12-item survey in which Patients are asked to reflect on their pain and functional ability over the previous 3 months There are two domains (pain and function) with six items or questions in each. Each item has four possible responses. In the scoring responses range from 0 to 4 where 0 represents the worst outcome and 4 represents the best. In this use, 48 is the maximum (and best) score achievable The scores for the 0-48 scale can be interpreted as follows Score 0 to 19 May indicate severe hip arthritis. Score 20 to 29 May indicate moderate to severe hip arthritis. Score 30 to 39 May indicate mild to moderate hip arthritis. Score 40 to 48 May indicate satisfactory joint function

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* A sufficient level of education to understand study procedures and be able to communicate with site personnel
* 50 eligible cases from the patients who underwent THA between December 2021 and December 2022 in our Assiut University Orthopaedics and Trauma surgery Department
* All ages of the patients
* All types of THA

Exclusion Criteria:

* Post traumatic Patients who are not available for 3 months follow-up
* Patients who refuse to participate in the study
* Rheumatoid arthritis
* All types of bone tumors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A dedicated sheet will be used to record patients' data . We conduct retrospective study.All patients followed and evaluated in our outpatient clinic at 3 month post-operatively. The questionnaire :(1) general satisfaction level after THA.(2) satisfaction level for 16 subordinate items : pain relief, walking on a flat surface , ascending stairs , getting in/out of cars, squatting, rising after squatting, putting on and tying shoes, walking fast or jogging, LLD, hip squeaking( cases of ceramic and non ceramic implant) , hip stiffness, abnormal feeling in the hip, muscle weakness when walking, hip numbness and discomfort in cold weather. The Harris Hip Scale (HHS) and Oxford Hip Score were developed for the assessment of the results of hip surgery such as THA
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction after Primary THA In Assiut University Hospitals | Baseline
  Percentage of improvement and satisfaction following THA during the follow up visits by using The Harris Hip Score which used as a measure of dysfunction so the higher the score, the better the outcome for the individual. The maximum score possible100 so results less than 80= dissatisfied group more than 80= satisfied group
measuring the level of satisfaction in primary cases of total hip arhroplasty | Baseline
  Percentage of improvement and level of satisfaction following THA by using Oxford Hip Score which used as a measure designed to assess disability in patients undergoing total hip arthroplasty. the maximum score is possible 48 so the higher results, the better outcome

SECONDARY OUTCOMES:
Percentage of improvement and clinical and functional outcome after total hip Arthroplasty | Baseline
  measuring the clinical and functional outcome at each visit by using
  The questionnaire that includes three majors parts
  (1) general satisfaction level after total hip arthroplasty .(2) satisfaction level for 16 subordinate items : pain relief, walking on a flat surface , ascending stairs , getting in/out of cars, squatting, rising after squatting, putting on and tying shoes, walking fast or jogging, (LLD) , hip squeaking( cases of ceramic and non ceramic implant) , hip stiffness, abnormal feeling in the hip, muscle weakness when walking, hip numbness and discomfort in cold weather(3) Ranking the top 5 important functions or issues among the 16 items , with "important" being defined as what patients are currently most concerned with

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okafor L, Chen AF. Patient satisfaction and total hip arthroplasty: a review. Arthroplasty. 2019 Sep 2;1(1):6. doi: 10.1186/s42836-019-0007-3. PMID 35240763
- [Background] Mancuso CA, Jout J, Salvati EA, Sculco TP. Fulfillment of patients' expectations for total hip arthroplasty. J Bone Joint Surg Am. 2009 Sep;91(9):2073-8. doi: 10.2106/JBJS.H.01802. PMID 19723982